CLINICAL TRIAL: NCT02085486
Title: Ultrasound Assisted Puncture of AV Fistulas in Chronic Hemodialysis Patients After a Short Learning Program in Bed-side Ultrasound for Hemodialysis Nurses by an Index Nurse - an Outcome Study
Brief Title: Ultrasound Assisted Puncture of AV Fistulas in Chronic Hemodialysis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of scientific interest
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SNCTP000000515
Record Dates: First submitted 2014-03-03; First posted 2014-03-12 (Estimated); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Dialysis; Fistula
Keywords: dialysis; av shunt; cannulation; ultrasound; outcome
MeSH Terms: conditions — Fistula; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-assisted puncture (Experimental): Ultrasound-assisted puncture by the nursing staff of patients with difficult AV-shunts.
  Interventions: Device: Ultrasound-assisted puncture
- Standard (Other): Classical method wtih inspection and palpation
  Interventions: Other: Standard

INTERVENTIONS:
Device: Ultrasound-assisted puncture — Portable ultrasound device
  Arms: Ultrasound-assisted puncture
Other: Standard — Standard inspection, palpation.
  Arms: Standard

SUMMARY:
The puncture of the vascular access in hemodialysis patients remains challenging even in the hands of experienced dialysis nurses. Unsuccessful punctures are associated with resource wastage, traumatism of the AV shunts, shortening of the effective dialysis time and poor patient satisfaction.

The use of ultrasound by emergency department nurses and technicians without prior ultrasound experience in patients with difficult intravenous access showed in several studies to be very efficient. The investigators expect to achieve similar results in cannulation of AV shunts by the dialysis nurse staff after a short learning program.

To show this, the investigators aim to conduct a trail where standard cannulation technique (inspection, palpation) will be compared with the ultrasound-assisted method in terms of efficacy, safety and patient satisfaction.

DETAILED DESCRIPTION:
Background

The vascular access plays a central role in patients with end-stage renal disease undergoing chronic hemodialysis. It is well documented from various previous studies that the confection of the dialysis access and subsequent complications represent a major cause of morbidity, hospitalization and additional costs in chronic dialysis patients.

In European countries most patients undergoing chronic hemodialysis use an arterio-venous fistula as permanent vascular access. Because of the anatomical differences of each individual and the accompanying chronic diseases affecting patients' vessels, cannulation of arterio-venous fistulas can be very challenging for the nursing personal and puncture failures necessitating repeated attempts are not so rare. The latter are often time-consuming and result in a loss of effective dialysis' time and reduced proceeded total blood volume, are associated with a higher rate of local complications due to repeated traumatisms of the vascular wall and can lead to severe pain with reduced patient satisfaction.

In the investigators' dialysis unit, when a dialysis nurse is not able to puncture a fistula she refers to an experienced nurse who tries to cannulate the fistula after thorough visual and palpatory evaluation. In case of another failure, the nursing team refers to the dialysis physician, who performs a short diagnostic bed-side ultrasound of the vascular access to rule out the presence of thrombosis or large hematoma. Using ultrasound-guidance provided by the physician or after being informed about the localization and depth of the ideal puncture site, the dialysis nurse tries then to puncture the fistula again. This often leads to a greater loss of time with reduced effective dialysis dose, increased need for human resources and low patient satisfaction.

The use of ultrasound by emergency department nurses and technicians without prior ultrasound experience in patients with difficult intravenous access showed in several studies to be very efficient. The method was safe, the procedure rapid, the patients more satisfied, the success rate as high as this from ultrasound trained emergency physicians and the need for physician intervention reduced. The achievement of similar results in AV fistula cannulation in hemodialysis patients would be very suitable.

The use of ultrasound in patients with recognized difficult fistulas by dialysis nurses after a short ultrasound learning program provided by an index nurse will enable to achieve a higher rate of satisfactory double-needle punctures, usual blood flow rates and full dialysis length with less time loss and increased patient satisfaction.

With this study prospective, single-centre, randomized, controlled study the investigators aim to show that the use of ultrasound by dialysis nurses in patients with difficult fistulas makes the punction of the fistulas easier than when assessing the fistula visually and manually.

Objective

The use of ultrasound in patients with recognized difficult fistulas by dialysis nurses after a short ultrasound learning program provided by an index nurse will enable to achieve a higher rate of satisfactory double-needle punctures, usual blood flow rates and full dialysis length with less time loss and increased patient satisfaction. With a prospective, controlled trail the investigators want to demonstrate this hypothesis.

Methods

A portable ultrasound device will be used by the nursing staff after a short learning program. Precise location of AV shunt segments and depth will be assessed in the case of a difficult shunt. This procedure will be compared with the standard inspection and palpation method.

ELIGIBILITY:
Inclusion Criteria:

* Forearm or upper arm AV-shunt (native, mixed, graft)
* Patients with recognized difficult vascular access at any time (potentially each patient)
* Written informed consent

Exclusion Criteria

* Recent AV-shunt surgery (< 48 h)
* Presence of large bandages or severe skin lesions in the area of interest
* Inability to understand the aim of the study and to give a written informed consent
* Single needle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Rate of successful cannulations of an AV-fistula | Immediately after the cannulation, expected to be after 10 minutes on average
  Satisfactory puncture of the fistula defined as the ability to achieve a full length dialysis (max. 10% reduction of the usual dialysis time), double-needle, and the usual blood flow rate (max. 15% reduction of the usual blood flow)

SECONDARY OUTCOMES:
Effective dialysis time | Directly after the treatment, expected to be after 3 to 4.5 hours
  Measured in minutes
Processed volume | Directly after the treatment, expected to be after 3 to 4.5 hours
Number of patients with late complications | At the following dialysis session, expected to be after 2-3 days
Patient satisfaction | Immediately after the canulation, expected to be after 10 minutes on average, and at the following dialysis session, expected to be after 2-3 days
  Measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kalicki, MD, Principal Investigator — Universitätsklinik für Nephrologie, Hypertonie und Klinische Pharmakologie, Inselspital Bern

REFERENCES:
- [Background] Feldman HI, Kobrin S, Wasserstein A. Hemodialysis vascular access morbidity. J Am Soc Nephrol. 1996 Apr;7(4):523-35. doi: 10.1681/ASN.V74523. PMID 8724885
- [Background] Hakim R, Himmelfarb J. Hemodialysis access failure: a call to action. Kidney Int. 1998 Oct;54(4):1029-40. doi: 10.1046/j.1523-1755.1998.00122.x. PMID 9767519
- [Background] Saudan P, Kossovsky M, Halabi G, Martin PY, Perneger TV; Western Switzerland Dialysis Study Group. Quality of care and survival of haemodialysed patients in western Switzerland. Nephrol Dial Transplant. 2008 Jun;23(6):1975-81. doi: 10.1093/ndt/gfm915. Epub 2007 Dec 22. PMID 18156654
- [Background] Brannam L, Blaivas M, Lyon M, Flake M. Emergency nurses' utilization of ultrasound guidance for placement of peripheral intravenous lines in difficult-access patients. Acad Emerg Med. 2004 Dec;11(12):1361-3. doi: 10.1197/j.aem.2004.08.027. PMID 15576530
- [Background] Bauman M, Braude D, Crandall C. Ultrasound-guidance vs. standard technique in difficult vascular access patients by ED technicians. Am J Emerg Med. 2009 Feb;27(2):135-40. doi: 10.1016/j.ajem.2008.02.005. PMID 19371518